CLINICAL TRIAL: NCT06966297
Title: Study of Calf Muscle Perfusion in Patients With Peripheral Arterial Disease After Revascularization Procedure Using Multispectral Optoacoustic Tomography
Brief Title: MSOT_PI Analysis of Revascularization Procedure Using Optoacoustic Imaging
Acronym: MSOT_PI
Status: Completed | Type: Observational
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Ulrich Rother, Senior Physician, University Hospital Erlangen
Other Study IDs: MSOT_PI
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: PAD; Vascular Diseases
Keywords: PAD; Optoacoustic Imaging
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- PAD Fontaine stage II endo: Patients in PAD Stage II receiving endovascular revascularization procedures
- PAD Fontaine stage II open: Patients in PAD Stage II receiving open surgical revascularization procedures
  Interventions: Diagnostic Test: Multispectral optoacoustic tomography
- PAD CLTI endo: Patients in PAD-CLTI (Chronic limb threatening ischemia) receiving endovascular revascularization procedures
  Interventions: Diagnostic Test: Multispectral optoacoustic tomography
- PAD CLTI open: Patients in PAD PAD-CLTI (Chronic limb threatening ischemia) receiving open surgical revascularization procedures
  Interventions: Diagnostic Test: Multispectral optoacoustic tomography

INTERVENTIONS:
Diagnostic Test: Multispectral optoacoustic tomography — Measurement of calf muscle Perfusion via Multispectral optoacoustic Tomography
  Groups: PAD CLTI endo; PAD CLTI open; PAD Fontaine stage II open

SUMMARY:
The aim of the proposed study is to analyse the improvement of the calf muscle perfusion of patients with PAD Fontaine stage II and critical limb threatheaning ischemia (CLTI) after endovascular and surgical revascularization procedures using multispectral optoacoustic tomography (MSOT)

DETAILED DESCRIPTION:
Since 2021, the University Hospital Erlangen (department of pediatrics) disposes of a CE-certified multispectral optoacoustic tomograph (MSOT). Similar to sonography, the MSOT technology allows for non-invasive, quantitative imaging of the composition and also oxygenation of target tissues such as muscle.

Just like with conventional sonography, the MSOT transducer head is placed on the skin of the examined person above the target organ. But instead of sound waves, energy is applied to the tissue via flashes of laser light. This leads to constant changes of minimal expansions and contractions (thermoelastic expansion) of different tissue components or molecules. The same examination unit that sends in the laser flashes can also detect the emitted ultrasound waves. In the newly configured device (Acuity Echo, iThera Medical GmbH, Munich, CE-certified), an extended spectrum of laser light can be used, enabling among others the derivation of values corresponding to hemoglobin and its oxygenation levels. As hemoglobin concentration and oxygenation status are markers for perfusion, MSOT-based imaging of these parameters could be a highly sensitive and reliable method to analyze muscle perfusion.

These parameters have already been successfully measured, validated and reproduced in preliminary studies. Furthermore, a first internal study (MSOT_PAD, NCT04641091) confirmed the hypothesis that data collected via MSOT can be used for PAD diagnostics. The derived concentration of oxygenated hemoglobin (HbO2) proved to be the most suitable measurement parameter. Correlations could be established between the measured HbO2 concentration and the radiological and clinical severity of the PAD.

These results are very promising in terms of using the MSOT technique in diagnosis and monitoring of PAD. In particular, the establishment of this method would be of great value for the examination of PAD patients in whom, due to previous illness such as severe chronic renal insufficiency or diabetes mellitus, the measurement of the ABI or the CCDS examination do not provide valid results due to progressive stiffening of the vascular wall (Mönckeberg mediasclerosis). This also applies to patients who, due to previous illness or operations, cannot perform treadmill exercise to determine the absolute walking distance. With MSOT, an objectifiable measurement method for non-invasive monitoring of the actual target organ muscle could be established for the first time, which would be especially helpful in the mentioned patient groups. Up until now there are no non-invasive measurement methods other than MSOT that can make transcutaneous statements about muscle perfusion.

In the previous study (MSOT_PAD, NCT04641091), differentiability of clinical PAD stages improved after a standardized exercise of a walking distance of 150 meters, with patients in the stage of intermittent claudication (IC, Fontaine stage II) being harder to differentiate compared to patients in stage III and IV. For diagnostic methods that address macrocirculation (especially ABI and FKDS), provocation tests are routinely used in PAD diagnostics and already standardized. As a rule, patients with PAD are stressed up to their personal stress limit (ischemia pain). The respective examination is then repeated afterwards. This increases the ability to differentiate macrocirculatory variables, especially for minor pathologies. We assume that this also applies to the hemoglobin concentrations (at the microcirculation level), even though up until now there are no measurement methods for this.

The MSOT technique, with its non-invasive, direct measurement of muscle perfusion, could prove to be particularly helpful for IC patients in terms of early diagnosis and follow-up. Where previously conservative therapy monitoring was based mainly on anamnesis, the MSOT technique could enable objective control and evaluation of the conservative and interventional/surgical treatment approaches. In the future this might entail further comparative outcome studies which might then even result in indication changes for the various therapeutic measures - which would improve the overall care situation of PAD patients.

In a further cross-sectional study, a large group of IC patients was examined using a more suited exercising of the calf muscle namely repeated heel raises until the occurrence of claudication pain. With this improved protocol, sensitivity and specificity of the procedure could be improved compared to the preliminary study.

With the help of this improved protocol we now want to examine whether and how the improved blood flow situation translates to the measured MSOT parameters. MSOT-scans of patients with PAD fontaine stage II and critical limb threathening ischemia will be conducted before and after endovascular or surgical revascularization procedure. . This comparison of muscle perfusion before and after revascularization is the obvious next step in this area of research. The study could help validate the therapeutic succes of said interventions as the currently available non-invasive diagnostics still pose limitations to objectively quantify the success of revascularization procedures.

As an additional target variable, the PAD-specific quality of life will be recorded via the VASCUQOL-6 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PAD confirmed by clinical examination and ABI (ABI ≤ 0.90)
* Planned for elective revascularization therapy
* Able to provide informed consent
* PAD stages II-IV Fontaine
* Age of > 18 years

Exclusion Criteria:

* Severe comorbid conditions

  * Non-PAD related walking impairments (e.g., neurological disorders)
  * Inability to comply with study protocols
  * PAD stage I
  * Age of < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 patients diagnosed with PAD were recruited for the study. Patients were included if they were scheduled for revascularization, either through endovascular therapy or an open surgical procedure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin associated parameters measured via Multispectral optoacoustic Tomography | 1 Hour

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larsen ASF, Reiersen AT, Jacobsen MB, Klow NE, Nordanstig J, Morgan M, Wesche J. Validation of the Vascular quality of life questionnaire - 6 for clinical use in patients with lower limb peripheral arterial disease. Health Qual Life Outcomes. 2017 Sep 22;15(1):184. doi: 10.1186/s12955-017-0760-3. PMID 28938901
- [Background] Lawall, H., P. Huppert, and G. Rümenapf. "S3-Leitlinie zur Diagnostik, Therapie und Nachsorge der peripheren arteriellen Verschlusskrankheit." Deutsche Gesellschaft für Angiologie und Deutsche Gesellschaft für Gefäßmedizin 30 (2015).
- [Background] Lanzer, P. (2018). Primary media sclerosis Mönckeberg: Diagnostic criteria. Cor et Vasa, 60(2), e205-e208.
- [Background] Alpert JS, Larsen OA, Lassen NA. Exercise and intermittent claudication. Blood flow in the calf muscle during walking studied by the xenon-133 clearance method. Circulation. 1969 Mar;39(3):353-9. doi: 10.1161/01.cir.39.3.353. No abstract available. PMID 4885945
- [Background] Karlas A, Masthoff M, Kallmayer M, Helfen A, Bariotakis M, Fasoula NA, Schafers M, Seidensticker M, Eckstein HH, Ntziachristos V, Wildgruber M. Multispectral optoacoustic tomography of peripheral arterial disease based on muscle hemoglobin gradients-a pilot clinical study. Ann Transl Med. 2021 Jan;9(1):36. doi: 10.21037/atm-20-3321. PMID 33553329